CLINICAL TRIAL: NCT07128108
Title: Multicenter Clinical Study on Noninvasive Assessment of Hepatic Steatosis and Fibrosis Using Visual Transient Elastography
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shenzhen Mindray Bio-Medical Electronics Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: Hepatus-V1
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Liver Injury; Mindray Hepatus 9 Ultrasound Diagnostic System
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Visual Transient Elastography (ViTE) Examination — Post-marketing product (Mindray Hepatus 9 Ultrasound Diagnostic System) for visual transient elastography examination in patients with liver injury.

SUMMARY:
Using liver biopsy as the gold standard, this study will conduct visual transient elastography (ViTE) examinations using Mindray Hepatus 9 ultrasound diagnostic system in patients with liver injury to evaluate the diagnostic efficacy of Liver Steatosis Analysis (LiSA) and ViTE for grading hepatic steatosis and fibrosis, and establish corresponding diagnostic thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18-65 years.
* Documented liver injury of any etiology with a liver biopsy performed within the past 2 weeks.
* Willing to undergo Visual Transient Elastography (ViTE) examination using Mindray Hepatus 9 Ultrasound System and capable of providing written informed consent.

Exclusion Criteria:

* Acute viral hepatitis.
* Right heart failure with either:Serum transaminases >5× upper limit of normal (ULN),Total bilirubin >85.5 μmol/L.
* History of hepatocellular carcinoma (HCC).
* Pregnancy.
* Patients with implantable medical devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver injury
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of LiSA and ViTE was evaluated using the area under the receiver operating characteristic curve (AUROC). | baseline
  Optimal cutoff values for LiSA and ViTE were determined by maximizing the Youden index, sensitivity (Se), and specificity (Sp). For each cutoff value, the following metrics with 95% confidence intervals (CI) were calculated: sensitivity (Se), specificity (Sp), positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Locations (1):
- XinHua Hospital Affiliated To Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No